CLINICAL TRIAL: NCT02991339
Title: The Effects of Dexamethasone Administration on Jaundice Following Liver Resection: a Randomized Controlled Trial
Brief Title: The Effects of Dexamethasone Administration on Jaundice Following Liver Resection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Deputy Director of the Department of Liver Surgery, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZS-SHC-DAJ
Record Dates: First submitted 2016-11-25; First posted 2016-12-13 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Liver Dysfunction; Hepatectomy; Bilirubinaemia; Jaundice
Keywords: Dexamethasone; Liver Dysfunction; Hepatectomy; Bilirubinaemia; Jaundice
MeSH Terms: conditions — Liver Diseases; Hyperbilirubinemia; Jaundice | interventions — Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 10 mg iv on day 1 and day 2, then 5 mg iv on day 3. For the patients the serum total bilirubin did not decrease to 1.5 ULN, then 5 mg iv on day 4.
  Interventions: Drug: Dexamethasone
- control (No Intervention): Patients are not treated with glucocorticoids.

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10 mg iv for 2 days; then 5 mg iv for 1 day
  Other Names: Dexamethasone Sodium Phosphate Injection
  Arms: Dexamethasone

SUMMARY:
The investigators were aiming to evaluate whether dexamethasone administration accelerates the recovery from hepatectomy-related jaundice and decreases the rates of post-hepatectomy liver failure and its safety in the subjects who developed elevated serum total bilirubin.

DETAILED DESCRIPTION:
Post-operative jaundice is one of the most common complications after hepatectomy for various liver tumors. Glucocorticoids, including dexamethasone, prednisolone, and methylprednisolone, were widely used to treat jaundice in the patients with severe hepatitis, liver dysfunction or liver failure. It was reported that glucocorticoids decrease the rates of liver dysfunction or mortality in those patients. However, whether post-operative glucocorticoids administration alleviated jaundice or deceased the rates of post-hepatectomy liver failure (PLF) yet to be determined. In this study, the investigators were aiming to evaluate whether dexamethasone administration accelerates the recovery from hepatectomy-related jaundice and decreases the rates of PLF and its safety in the subjects who developed elevated serum TB.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent open hepatectomy for liver tumors
* Preoperative liver function was Child-Pugh A, and the liver shear wave elastography (SWE) < 30 kPa
* Postoperative serum total bilirubin > 2.5 ULN in 7 days after hepatectomy

Exclusion Criteria:

* Patients with hilar cholangiocarcinoma or other disease with obstructive jaundice
* Complicating disease with severe dysfunction in respiratory or circulation system or kidney.
* Patients with contraindication of glucocorticoids, including severe infection, active GI bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
period in days from the day serum total bilirubin (TB) >=2.5 ULN to the day TB decreased to 1.5 ULN | up to 30 days after hepatectomy

SECONDARY OUTCOMES:
The dynamic change of serum total bilirubin | up to 30 days after hepatectomy
length of hospital stay | up to 30 days after surgery
inhospital expenses | up to 30 days after surgery
post-operative complications, including postoperative liver failure, infection and GI bleeding | up to 30 days after surgery
The dynamic change of serum glutamine aminotransferase | up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Sun, MD, Principal Investigator — Liver Cancer Insitute and Zhongshan Hospital, Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Result] Mathurin P, O'Grady J, Carithers RL, Phillips M, Louvet A, Mendenhall CL, Ramond MJ, Naveau S, Maddrey WC, Morgan TR. Corticosteroids improve short-term survival in patients with severe alcoholic hepatitis: meta-analysis of individual patient data. Gut. 2011 Feb;60(2):255-60. doi: 10.1136/gut.2010.224097. Epub 2010 Oct 12. PMID 20940288
- [Result] Thursz MR, Forrest EH, Ryder S; STOPAH investigators. Prednisolone or Pentoxifylline for Alcoholic Hepatitis. N Engl J Med. 2015 Jul 16;373(3):282-3. doi: 10.1056/NEJMc1506342. No abstract available. PMID 26176387
- [Result] Chen JF, Wang KW, Zhang SQ, Lei ZY, Xie JQ, Zhu JY, Weng WZ, Gao ZL, Lin BL. Dexamethasone in outcome of patients with hepatitis B virus-related acute-on-chronic liver failure. J Gastroenterol Hepatol. 2014 Apr;29(4):800-6. doi: 10.1111/jgh.12454. PMID 24224656
- [Result] Yamashita Y, Shimada M, Hamatsu T, Rikimaru T, Tanaka S, Shirabe K, Sugimachi K. Effects of preoperative steroid administration on surgical stress in hepatic resection: prospective randomized trial. Arch Surg. 2001 Mar;136(3):328-33. doi: 10.1001/archsurg.136.3.328. PMID 11231856